CLINICAL TRIAL: NCT05121636
Title: Clinical Outcomes Following Total Joint Replacement With Corin Prostheses : Trinity™ Cup and MetaFix™ Collared Stem
Brief Title: Clinical Outcomes Following Total Joint Replacement With Corin Prostheses: Corin MetaFix Collared Stem
Status: Active, not recruiting | Type: Observational
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP2016-01
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: MetaFix Collared Stem — Patients received the MetaFix Collared stem during there Total Hip Arthroplasty

SUMMARY:
Assessment of the clinical performance and survivorship of the Corin Total Hip System with Trinity™ cup MetaFix™ Collared stem in a prospective study. The primary endpoint of the study is to evaluate the 3-year survivorship and clinical performance of the Corin Total Hip System using Trinity™ cup and MetaFix™ Collared stem. Additionally, the study follow up will continue until 10 years for subjects who consent to do.

DETAILED DESCRIPTION:
The primary objective is the 3-year survivorship of the study devices.

The Secondary Objectives include:

* The improvement of clinical outcomes:

  * Oxford Hip Score (OHS) up to 10-year follow-up
  * Harris Hip Score (HHS) up to 10-year follow-up
  * Hip disability and Osteoarthritis Outcome Score (HOOS) up to 10-year follow-up
* Safety performance monitoring including hip- and device-related AEs and the revision rate up to 10-year follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring a THR

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring a THR were identified and screened according to the Indications for use and the contraindications for implantation of the MetaFix™ collared femoral stem and the Trinity™ acetabular cup were invited to consent to the study. No specific exclusion criteria were defined for this study.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-06-12 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2027-09-02 (Estimated)

PRIMARY OUTCOMES:
Post operative survivorship of MetaFix Collared Stem at 3-year follow-up | 3 years
  Survivorship measured via Kaplan-Meier (KM) curve.

SECONDARY OUTCOMES:
Harris Hip Score (HHS) up to 10-year follow-up | Baseline to 10 years
  Harris Hip Score is a disease-specific scoring system, originally intended as an outcome score after arthroplasty surgeries that includes the domains of function, pain, motion and deformity. Minimum score is 0, Maximum score is 100. The score is reported as 90-100 for excellent results, 80-89 for good, 70-79 for fair, 60-69 for poor, and below 60 for a failed result.
Oxford Hip Score (OHS) up to 10-year follow-up | Baseline to 10 years
  Oxford Hip Score is a patient-centered questionnaire that is designed to assess functional ability and pain from the patient's perspective. It is a short, twelve-item questionnaire developed for completion by patients undergoing THA. Minimum score 0 indicating worst outcome, maximum score 48 indicating best outcome.
Hip disability and Osteoarthritis Outcome Score (HOOS) up to 10-year follow-up | Baseline to 10 years
  The validated Hip disability and Osteoarthritis Outcome Score questionnaire is designed for patients with hip Osteoarthritis, it consists of 40 questions which assesses Pain, Symptoms, Activities of Daily Living, Sport and Recreational and Hip related Quality of life. To answer the questions, standardized answer options are given in 5 Likert-boxes with scores from 0 to 4 (no, mild, moderate, severe and extreme).
  To interpret the score, the outcome measure is transformed in a worst to best scale from 0 to 100, with 100 indicating no symptoms and 0 indicating extreme symptoms.
Hip- and device-related adverse events up to 10-year follow-up | Baseline to 10 years
  All hip-related and device-related complications, including those occurring during the surgical procedure and throughout the postoperative evaluations, are required to be documented and reviewed
Post operative survivorship of MetaFix Collared Stem at 10-year follow-up | Baseline to 10 years
  Survivorship measured via Kaplan-Meier (KM) curve.
MetaFix Collared Stem radiographic performance up to 10-years | Baseline to 10 years
  Radiographic assessment considering radiolucent lines, stem alignment, heterotopic ossifications, osteolysis.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Barnett, Principal Investigator — Hoag Orthopedic Institute

IPD SHARING:
Plan to Share IPD: Undecided